CLINICAL TRIAL: NCT06420687
Title: The Functional Importance of Powered Wrist Flexion for Transradial Prosthetic Users
Brief Title: GaMA Metric to Quantify Functional Importance of Various Upper Limb Prosthetic Devices
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: University of Alberta (Other)
Responsible Party: Principal Investigator, Laura Miller, Team Scientist III, Shirley Ryan AbilityLab
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: STU00211352
Record Dates: First submitted 2024-05-13; First posted 2024-05-20 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Amputation; Amputation, Traumatic; Amputation; Traumatic, Hand; Amputation; Traumatic, Limb
Keywords: Upper Limb Prosthetic Users
MeSH Terms: conditions — Amputation, Traumatic

STUDY DESIGN:
Intervention Model Description: The GaMA metric will utilize motion capture and eye tracking hardware and software during the administration of functional tasks while research participants are using commercially available prosthetic devices and investigational prosthetic devices currently in development.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Able-bodied participants (No Intervention): Participants without amputation were enrolled to collect normative data for system validation. Adhesive motion capture markers will be placed on both arms (upper arm, forearm, hand and finger tips), thoracic spine and sacrum. The participant wears a specialized headband/glasses with an attached camera for eye tracking. The participant will pick up and move objects of different shapes to and from various heights.
- Transradial amputee participants (Active Comparator): Individuals using their home prosthesis when available. Adhesive motion capture markers will be placed on both arms (upper arm, forearm, hand and finger tips), thoracic spine and sacrum. The participant will wear a headband with attached markers for eye tracking. The participant will pick up and move objects of different shapes to and from various heights.
  Interventions: Device: Clinically prescribed prosthesis
- Transradial amputee participants - Wrist rotation+1 dof hand (Experimental): Individuals with transradial amputation fit with experimental prosthesis consisting of wrist rotation and one degree of freedom hand. Adhesive motion capture markers will be placed on both arms (upper arm, forearm, hand and finger tips), thoracic spine and sacrum. The participant will wear a headband with attached markers for eye tracking. The participant will pick up and move objects of different shapes to and from various heights.
  Interventions: Device: Experimental prosthesis - Wrist rotation + 1-DOF
- Transradial amputee participants - Wrist rotation + wrist flexion +1 dof hand (Experimental): Individuals with transradial amputation fit with experimental prosthesis consisting of wrist rotation, wrist flexion and one degree of freedom hand. Adhesive motion capture markers will be placed on both arms (upper arm, forearm, hand and finger tips), thoracic spine and sacrum. The participant will wear a headband with attached markers for eye tracking. The participant will pick up and move objects of different shapes to and from various heights.
  Interventions: Device: Experimental prosthesis - Wrist rotation + Wrist flexion +1-DOF
- Transradial amputee participants - Wrist rotation + multi degree freedom hand (Experimental): Individuals with transradial amputation fit with experimental prosthesis consisting of wrist rotation and multi degree freedom hand. Adhesive motion capture markers will be placed on both arms (upper arm, forearm, hand and finger tips), thoracic spine and sacrum. The participant will wear a headband with attached markers for eye tracking. The participant will pick up and move objects of different shapes to and from various heights.
  Interventions: Device: Experimental prosthesis - Wrist rotation + Multi DOF hand
- Transradial amputee participants - Wrist rotation + wrist flexion + multi degree freedom hand (Experimental): Individuals with transradial amputation fit with experimental prosthesis consisting of wrist rotation, wrist flexion and multi degree freedom hand. Adhesive motion capture markers will be placed on both arms (upper arm, forearm, hand and finger tips), thoracic spine and sacrum. The participant will wear a headband with attached markers for eye tracking. The participant will pick up and move objects of different shapes to and from various heights.
  Interventions: Device: Experimental prosthesis - Wrist rotation + wrist flexion + Multi DOF hand

INTERVENTIONS:
Device: Clinically prescribed prosthesis — Clinically prescribed prosthesis:
  Arms: Transradial amputee participants
Device: Experimental prosthesis - Wrist rotation + 1-DOF — 1-DOF wrist rotation and1-DOF hand
  Arms: Transradial amputee participants - Wrist rotation+1 dof hand
Device: Experimental prosthesis - Wrist rotation + Wrist flexion +1-DOF — 2-DOF wrist (rotation and flexion) and 1-DOF hand
  Arms: Transradial amputee participants - Wrist rotation + wrist flexion +1 dof hand
Device: Experimental prosthesis - Wrist rotation + Multi DOF hand — 1-DOF wrist rotation and multi-DOF hand
  Arms: Transradial amputee participants - Wrist rotation + multi degree freedom hand
Device: Experimental prosthesis - Wrist rotation + wrist flexion + Multi DOF hand — 2-DOF wrist (rotation and flexion) and multi-DOF hand
  Arms: Transradial amputee participants - Wrist rotation + wrist flexion + multi degree freedom hand

SUMMARY:
The goal of this study is to utilize the Gaze and Movement Assessment (GaMA) metric to assess the effect of different prosthetic components on compensatory movements used to complete activities of daily living.

DETAILED DESCRIPTION:
Evaluating the benefit of new prosthetic components and control mechanisms can be challenging, as most validated outcome measures assess the time required to complete various tasks without assessing the quality of the movement or the specific DOF(s) activated to accomplish the task. There are no adequate methods to evaluate the impact of new technology. The functional outcome measures recommended by The Academy of Prosthetics and Orthotics Upper Limb Prosthetic Outcome Measures (ULPOM) committee, which provided recommendations for measuring functional effectiveness of prosthetic treatment, mainly focus on the time to complete the task rather than assessing the compensatory movements.

The Gaze and Movement Assessment (GaMA) is a new validated and standardized metric to quantify the functional characteristics of prosthesis use by quantifying motion (three dimensional angular kinematics), gaze behavior and performance during simulated real-world tasks. There are two tasks, the Cup Transfer Task and the Pasta Box Task, used with the GAMA testing hardware. The tasks require movements representing day-to-day functional requirements, while challenging typical prosthetic limitations such as reaching and transporting objects at varying heights and across the body and lack of wrist motion. Each task can be subdivided into specific phases of reaching, grasping, transporting and releasing objects. A performance aspect encourages the participant to work efficiently, and tasks are short to allow multiple repetitions within a reasonable testing time frame to assess performance consistency. By breaking down each task into movements (i.e., of the pasta box from one shelf to the next), and each movement into specific phases (reach, grasp, transport, and release), the investigators can examine these components individually. It is hypothesized that additional degrees-of-freedom (for example wrist flexion) may require more time but will reduce the compensatory movements required to complete the tasks.

The primary endpoint of the study is to quantify the effect of various prosthetics components on kinematics.

The secondary endpoint is to obtain normative data for the GaMA system and system validation.

ELIGIBILITY:
Inclusion Criteria:

* A unilateral upper limb amputation or absence below the elbow
* Ability to use a myoelectric prosthesis
* English Speaking

Exclusion Criteria:

* Significant new injury that would prevent use of a prosthesis: The ability to consistently wear a prosthesis and perform activities of daily living and specific performance tasks is necessary to evaluate the relative benefits of the interventions.
* Cognitive impairment sufficient to adversely affect understanding of or compliance with study requirements, ability to communicate experiences, or ability to give informed consent: The ability to understand and comply with requirements of the study is essential in order for the study to generate useable, reliable data.
* Significant other comorbidity: Any other medical issues or injuries that would preclude completion of the study, use of the prostheses, or that would otherwise prevent acquisition of useable data by researchers

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-04-20 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Kinematics data while performing the Pasta Box Task | After 6-week home trial
  Utilizes motion capture hardware during prosthesis use and collects three dimensional angular kinematics, gaze behavior and performance during simulated tasks.
  Participants move a pasta box from the target on a side cart at the right side of the body onto a mid-height shelf target in front of them. Then they move the box from the mid-height shelf target to the high shelf target on the opposite side. Finally, they pick up the pasta box from the high shelf target and return it to the initial position.
  Each task can be subdivided into specific phases of reaching, grasping, transporting and releasing objects. By breaking down each task into movements, and each movement into specific phases (reach, grasp, transport, and release), the investigators can examine these components individually.
Kinematics data while performing the Cup Transfer Task | After 6-week home trial
  Utilizes motion capture hardware during prosthesis use and collects three dimensional angular kinematics, gaze behavior and performance during simulated tasks.
  The Cup transfer task consists of moving two cups filled with beads (simulating being filled with liquid) over a partition and back again for a total of four object movements. The cups are deformable and will spill beads if grabbed too hard. Like in the Pasta task, participants start each trial with their hand in the home position and their eyes fixated on a centered motion capture marker.
  Each task can be subdivided into specific phases of reaching, grasping, transporting and releasing objects. By breaking down each task into movements, and each movement into specific phases (reach, grasp, transport, and release), the investigators can examine these components individually.

SECONDARY OUTCOMES:
Eye gaze data while performing the Pasta Box Task | After 6 week home trial
  Eye tracking hardware during prosthesis use the GAMA collects three dimensional gaze behavior and performance during simulated tasks.
Eye gaze data while performing the Cup Transfer Task | After 6 week home trial
  Eye tracking hardware during prosthesis use the GAMA collects three dimensional gaze behavior and performance during simulated tasks.

CONTACTS AND LOCATIONS:
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States